CLINICAL TRIAL: NCT06770998
Title: A Prospective Randomized Study of a Novel EEG Neurofeedback System for the Treatment of PTSD Using Machine Learning-Based Amygdala Biomarkers
Brief Title: A Study of a Novel EEG Neurofeedback System for PTSD Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Atlanta Veterans Education and Research, Inc. (Other)
Collaborators: GrayMatters Health Ltd. (Industry); Rochester Institute of Technology (Other); NYU Langone Health (Other); Atlanta VA Medical Center (U.S. Federal Agency); Birmingham VA Health Care System (U.S. Federal Agency); Ralph H. Johnson VA Medical Center (U.S. Federal Agency); VA Boston Healthcare System (U.S. Federal Agency); CTP Inc (Unknown); BioStats Statistical Consulting Ltd (Unknown); ShareCRF (Unknown); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNC138; TP230099 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2024-12-19; First posted 2025-01-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-07

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: EEG; trauma; neurofeedback; biofeedback; stress disorders, traumatic; trauma and stressor related disorders; military trauma; civilian trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries; Stress Disorders, Traumatic; Trauma and Stressor Related Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prism training (Active Comparator)
  Interventions: Device: EEG-neurofeedback training
- Sham training (Sham Comparator)
  Interventions: Device: Sham training

INTERVENTIONS:
Device: EEG-neurofeedback training — 15 training sessions (twice/week) plus two booster training sessions added to treatment as usual.
  Other Names: Prism training; amyg-EFP training; active Prism training
  Arms: Prism training
Device: Sham training — 15 sham sessions (twice/week) plus two sham booster sessions added to treatment as usual.
  Other Names: sham Prism training
  Arms: Sham training

SUMMARY:
The goal of this clinical trial is to learn if training with the Prism system can reduce PTSD symptoms in US military Veterans and civilians with PTSD. Prism is a form of neurofeedback training that uses EEG signals to promote self-regulation of brain function. The main question this study aims to answer is:

Does Prism training lead to decreased PTSD symptoms in US Veterans and civilians when used in addition to usual PTSD treatment?

Researchers will compare Prism training to a sham training (a look-alike training that does not provide real feedback on brain activity) to see if Prism training decreases PTSD symptoms.

Participants will:

* Complete two one-hour in-person training sessions a week for about 8 weeks (15 sessions)
* Complete two booster training sessions one month and two months after finishing the main training course
* Participate in three detailed interviews: one before training, a second after nine weeks of training, and a third one month after the last booster training session (about 20 weeks after the initial visit)

ELIGIBILITY:
Inclusion Criteria

Subjects must meet the following inclusion criteria:

1. Ages 18 to 65 (older limit to avoid those with potentially reduced brain plasticity due to age);
2. Male, female, and gender-nonconforming subjects will be allowed. Sites will make efforts to enroll both male and female subjects in roughly equal proportions;
3. Diagnosis of PTSD comorbidities will be confirmed by clinical chart review and structured interview with the Diagnostic Interview for Anxiety, Mood, and Obsessive-compulsive and Related Neuropsychiatric Disorders (DIAMOND), a semi-structured diagnostic interview instrument for DSM-5 psychiatric disorders with good test-retest reliability (Tolin et al. 2018);
4. Diagnosis of PTSD based on CAPS-5-R (scored as CAPS-5) total score with a minimum severity score of 26 at Baseline in the CAPS-5 score;
5. 1-26 years from index trauma;
6. Ability to give signed informed consent according to the judgment of the site investigator;
7. Normal or corrected-to-normal vision of at least 20/30 as per eye chart screening;
8. Normal or corrected-to-normal hearing as per subject report and interview with study staff;
9. Willingness and ability to adhere to the study schedule;
10. Comorbid major depression will be allowed as long as the primary care is PTSD, because it is frequently comorbid with PTSD, and its inclusion will render our study results salient to the real-world clinical population;*
11. Any psychotropic medication must have been at a stable dose for at least 4 weeks prior to screening;
12. At the time of recruitment, patients must have no plan of changing their medication or psychotherapy during the study duration if applicable (subjects will only be dropped if significant psychotropic medication changes happen as a result of clinical instability that, in the opinion of the principal investigator (PI), would jeopardize their ability to learn or participate).

    * Note: This is a clarification that comorbid depression is allowed and not an inclusion requirement.

Exclusion Criteria

Potential subjects will be excluded for the following:

1. Completed at least one adequate course of trauma-focused behavioral therapy in the past one (1) year without improvement in PTSD symptoms, as documented in medical records. (Subjects are ineligible if medical records do not show evidence of symptom improvement from the previous trauma focused therapy that had been conducted in the year prior to Screening); Non-response will be determined by clinical judgment and qualitative note content. If PCL-5 or CAPS-5 scores are available within 2 weeks prior to beginning treatment and within 2 weeks post-treatment, an improvement of <10 points in PCL-5 and <10 points in CAPS-5 will be used as a threshold indicating non-response in addition to clinical judgement.

   • Note: This criterion is to avoid treatment resistant patients; such patients will be enrolled in future studies);
2. Lifetime diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar I or II disorder, psychosis not otherwise specified, or delusional disorder;
3. Any Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) Mood or anxiety disorder (in addition to those described in the previous exclusion) that is the primary focus of mental health treatment in the 6 months prior to screening, per the site investigator's clinical judgment;
4. Intellectual disability (known full scale IQ<70) per the site investigator's clinical judgment;
5. DSM-5 diagnosis of moderate or severe substance use disorder within 3 months of screening;
6. Prescribed benzodiazepine which cannot be stopped for the duration of the study (with a washout period of at least 2 weeks prior to the first Prism training session) or replaced with short-acting benzodiazepines taken only at night for sleeping;
7. Any suicidal behavior in the last 6 months (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior) prior to screening and during the screening period and or current (in the last 6 months) significant suicidality (defined as Level 4+ on the C-SSRS) or current significant homicidality;
8. Within 3 months of beginning cognitive behavioral therapy (CBT) or any evidence-based PTSD psychotherapy, although continuing established maintenance supportive therapy will be permitted;
9. Any significant neurological/neurosurgical history, including brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality or known cognitive impairment;
10. A history of moderate or severe traumatic brain injury (TBI) or history of gross structural damage on brain imaging;
11. Any unstable medical condition per the investigator's clinical judgment;
12. Any psychiatric hospitalization within the last 6 months;
13. Enrollment in another interventional clinical study at screening or within 2 months prior to screening, or within the duration of this study;
14. Pregnancy is allowed, but excluded if at week 20 or later in the pregnancy at Baseline because early labor in the late term of the pregnancy would require the subject to withdraw from the study.
15. Acute symptoms of infection with SARS-CoV-2 (COVID-19) at time of screening or 2 months prior to screening as per interview and chart review;
16. Under criminal investigation or pending legal charges with potential incarceration;
17. Individuals who lack stable contact information (including lack of a telephone number);
18. Subjects who anticipate working during the hours of midnight to 6 AM during the study;
19. Subjects with narcolepsy;
20. Subjects who have a Legally Authorized Representative;
21. A positive result on the urine toxicology screen for any illegal substance besides marijuana. * * Note: If urine tests positive for any illegal substance, the results will not be included in the subject's medical record. However, these test results will remain part of the subject's confidential study record.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Total CAPS-5-R score change from Baseline to Week 9 | From enrollment to the end of 8 weeks' training (twice per week)
  Participants will take the Clinician-Administered PTSD Scale for DSM-5 Revised (the CAPS-5-R) before beginning Prism training. The CAPS-5-R assesses PTSD symptom severity with total scores that range from 0-80, with higher scores indicating more severe symptoms. There are multiple ways to score the CAPS-5-R; this study will score the CAPS-5-R using the same 0-80 score range used on the CAPS-5 (the previous version of the same assessment) so that the results from this study can be more easily compared to results from previous studies on the Prism training system. Participants' scores on the CAPS-5-R after completing training will be compared to their pre-training scores to determine whether the Prism training group shows a greater reduction in PTSD symptoms than the Sham training group.

SECONDARY OUTCOMES:
Total CAPS-5-R score change from Baseline to Week 20 | From enrollment to 20 weeks (including an initial 8 weeks of biweekly training and two booster sessions at Week 12 and Week 16)
  Participants will take the Clinician-Administered PTSD Scale for DSM-5 Revised (the CAPS-5-R) before beginning Prism training. The CAPS-5-R assesses PTSD symptom severity with total scores that range from 0-80, with higher scores indicating more severe symptoms. There are multiple ways to score the CAPS-5-R; this study will score the CAPS-5-R using the same 0-80 score range used on the CAPS-5 (the previous version of the same assessment) so that the results from this study can be more easily compared to results from previous studies on the Prism training system. Scores on the CAPS-5-R at 20 weeks after the first assessment (about one month after the second booster session) will be compared to the baseline CAPS-5-R score to determine whether the changes due to Prism training in the Prism training group vs the Sham training group persist over time.

OTHER OUTCOMES:
Exploratory outcome: change in PCL-5 score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether PTSD symptoms as measured by the PTSD Checklist for DSM-5 (PCL-5) decrease from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The PCL-5 measures PTSD symptoms. Total scores range from 0-80, with higher scores representing more severe symptoms.
Exploratory outcome: change in ACPL score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether PTSD symptoms as measured by the Abbreviated PTSD Checklist for DSM-5 (APCL) decrease from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The ACPL measures PTSD symptoms. Total scores range from 0-16, with higher scores representing more severe symptoms.
Exploratory outcome: change in HAM-D score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether depressive symptoms as measured by the Hamilton Depression Inventory (HAM-D) decrease from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The HAM-D measures depression symptoms. Scores range from 0-66, with higher scores representing more severe symptoms.
Exploratory outcome: change in PHQ-9 scores from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether depressive symptoms as measured by the Patient Health Questionnaire (PHQ-9) decrease from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The PHQ-9 measures depression symptoms. Total scores range from 0-27, with higher scores representing more severe symptoms.
Exploratory outcome: change in STAI score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether anxiety symptoms as measured by the State-Trait Anxiety Inventory (STAI) decreases from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The STAI measures anxiety symptoms. Total scores range from 20-80, with higher scores representing more severe symptoms.
Exploratory outcome: change in GAD-7 score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether anxiety symptoms as measured by the Generalized Anxiety Disorder (GAD-7) scale decreases from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The GAD-7 measures anxiety symptoms. Total scores range from 0-21, with higher scores representing more severe symptoms.
Exploratory outcome: change in CGI responses from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Using the Clinical Global Impression Scale (CGI), determine whether general mental wellbeing improves in correspondence to treatment from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The CGI assesses severity of current illness (1-7 ranging from healthy to very ill), global improvement in response to treatment (1-7 ranging from significant improvement to significant worsening) and efficacy of treatment (describes the risk-to-benefit ratio of treatment).
Exploratory outcome: change in PSQI score from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether sleep quality as measured by the Pittsburgh Sleep Quality Index (PSQI) improves from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The PSQI measures sleep quality. Total scores range from 0-21, with higher scores representing more disturbed sleep.
Exploratory outcome: change in ERQ scores from Baseline to Week 9 and from Baseline to Week 20 | 20 weeks (assessed at Week 9 and Week 20)
  Determine whether emotion regulation as measured by the Emotion Regulation Questionnaire (ERQ) improves from Baseline to Week 9 and from Baseline to Week 20 in the Prism treatment group compared to the Sham treatment group. The ERQ measures emotion regulation in terms of Cognitive Reappraisal and Expressive Suppression. Cognitive Reappraisal scores range from 0-42, with higher scores indicating greater likeliness to regulate emotions through cognitive reframing. Expressive Suppression scores range from 0-28, with higher scores indicating more suppression of emotional expression.
Exploratory outcome: identifying subject groups who would benefit from changes in the Prism training structure | 20 weeks
  Conduct a comprehensive analysis, combining Prism data with subject demographics, symptom ratings, and concomitant treatment, to develop prediction models which will be validated and used to predict treatment response and personalize Prism treatments.
  Specific subject groups will be identified for whom the prediction engines can optimize Prism treatment based on patient characteristics. Using the algorithms developed, we will combine Prism-extracted data with clinical and demographic information to identify treatment regimen adjustments (e.g., treatment duration, time between sessions, and number of booster sessions) that may benefit specific patient groups.
  The large-scale Prism data, combined with validated clinical measurements and subject characteristics, will allow Prism treatment personalization by predicting individual treatment responses. This will lay the groundwork for optimizing combinations of pharmacological and non-pharmacological treatments.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Birmingham VA Medical Center, Birmingham, Alabama
  - Atlanta VA Medical Center, Decatur, Georgia
  - Boston VA Healthcare System, Boston, Massachusetts
  - New York University Grossman School of Medicine, New York, New York
  - University of Rochester Medical Center (URMC), Rochester, New York
  - Charleston VA Medical Center, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No